CLINICAL TRIAL: NCT02478112
Title: Multicentre Study Evaluating the Use of a Biodegradable Balloon for the Treatment of Prostate Cancer (of Intermediate Risk) by Intensity Modulated Conformal Radiotherapy (BioPro-RCMI)
Brief Title: Use of a Biodegradable Balloon for the Treatment of Prostate Cancer by Intensity Modulated Radiotherapy (BioPro-RCMI)
Acronym: BioPro-RCMI
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Aquilab SAS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BioPro-RCMI-1505; N° IdRCB : 2015-A01041-48 (Other: ANSM)
Record Dates: First submitted 2015-06-15; First posted 2015-06-23 (Estimated); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Prostate Cancer
Keywords: Intensity Modulated Radiotherapy; Balloon implant
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biodegradable Balloon Implant (Experimental): Biodegradable balloon implanted before radiotherapy
  Interventions: Device: Biodegradable balloon implant

INTERVENTIONS:
Device: Biodegradable balloon implant — Implantation under general anaesthesia of a biodegradable balloon before radiation therapy for prostate cancer
  Other Names: BioProtect Balloon Implant System

SUMMARY:
The benefit of dose escalation in radiotherapy (RT) for biochemical control of prostate cancer is a clearly established fact based on the results of different published prospective trials. This benefit, acquired with three-dimensional conformal radiation technique is counterbalanced by an increase in urinary and gastrointestinal toxicity. The joint progress of dose planning systems and multileaf collimators (MLC) technology have enabled the Intensity Modulated Radiation Therapy (IMRT). Recently the contribution of "spacers" positioned in the septum between the rectum and the prostate could improve the functional results of IMRT in terms of rectal toxicity.

The aim of the investigators study is to assess the dosimetric gain from the contribution of the implantable BioProtect balloon on organs at risk.

DETAILED DESCRIPTION:
Patients eligible for the trial and having signed their consent to participate will undergo a scan to verify the possibility of implantation of the balloon. Before and after implantation of the balloon, a dosimetric scan will be performed. Radiotherapy will be administered according to the habits of each centre : Intensity modulated radiotherapy : 2 Gy / session, 5 weekly sessions, total dose of 74-80 Gy (+/- associated with an hormone therapy).

Patients will have a clinical examination :

* prior to the start of treatment
* once a week during the radiotherapy
* at the end of the radiotherapy
* and at the end of the study.

They will also complete quality of life questionnaires :

* prior to the start of treatment
* at mid-treatment
* at the end of the radiotherapy
* and at 3, 6, 12 and 24 months after the end of the radiotherapy.

Finally, patients will undergo a laboratory examination :

* prior to the start of treatment
* 3 months after the end of the radiotherapy
* and then every 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over 18 years old
2. With a localized adenocarcinoma of the prostate

   * of intermediate risk of D'AMICO
   * and of stage MRI < T3
3. Requiring a treatment with Intensity Modulated Radiotherapy
4. PSA (Prostate-Specific Antigen) levels ≤ 20 ng/mL before external beam radiotherapy
5. Prostate volume > 15 cc
6. Short hormone therapy possibly associated (4-6 months)
7. Patient without clinical signs of progressive disease (Performing a bone scan and a CT scan is optional)
8. Performance status ECOG (Eastern Cooperative Oncology Group) ≤ 1
9. Life expectancy ≥ 10 years
10. Informed consent signed

Exclusion Criteria:

1. Incompatibility to the implantation of a Bioprotect balloon :

   * ongoing anticoagulant by vitamin K antagonist (VKA) or heparintherapy
   * patient with immunosuppression or with serious chronic diseases such as heart failure, cirrhosis, chronic kidney failure, colic or rectal digestive inflammatory disease
   * history of prostatitis or of lower gastrointestinal infection treated or ongoing
   * history of recto-colic inflammatory disease or of repeated prostatic resections
   * untreated perineal wound
2. Prior treatment with hormone therapy
3. History of another invasive cancer within 5 years prior to study entry (with the exception of a treated basal cell skin carcinoma)
4. History of pelvic radiotherapy
5. Severe hypertension non controlled by an adapted treatment (≥ 160 mm Hg in systole and/or ≥ 90 mm Hg in diastole)
6. Ongoing antineoplastic therapy
7. Person deprived of liberty or under tutorship
8. Inability to submit to the medical monitoring of the study for geographical, social or psychological reasons.
9. Conformal radiotherapy without intensity modulation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-11-25 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Dosimetric gain from the contribution of the balloon on organs at risk | 24 months
  Evaluation by comparison of the dosimetric scans performed before and after the implantation of the balloon.

SECONDARY OUTCOMES:
Urinary and rectal toxicity | 24 months
  Urinary and rectal toxicity evaluated according to NCI-CTCAE v4.0
Stages of the implantation of the Bioprotect balloon | 1 week
  Monitoring of the balloon by Cone Beam Computed Tomography during the radiotherapy.
Technical feasibility of the implantation of the Bioprotect balloon | 1 week
  Monitoring of the balloon by Cone Beam Computed Tomography during the radiotherapy.
Quality of life by QLQ-C30 | 24 months
  Quality of life measured by the QLQ-C30 questionnaire of the EORTC (European Organisation for Research and Treatment of Cancer) and by the QLQ-C30 PR25 module and the International Prostate Symptom Score (IPSS)

CONTACTS AND LOCATIONS:
Overall Officials: David PASQUIER, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (6):
- France (6):
  - Institut Bergonié, Bordeaux
  - Centre Léonard de Vinci, Dechy
  - Clinique Hartmann, Levallois-Perret
  - Centre Oscar Lambret, Lille
  - Centre de Cancérologie Paris Nord, Sarcelles
  - Clinique Pasteur, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pasquier D, Bogart E, Bonodeau F, Lacornerie T, Lartigau E, Latorzeff I. BioPro-RCMI-1505 trial: multicenter study evaluating the use of a biodegradable balloon for the treatment of intermediate risk prostate cancer by intensity modulated radiotherapy; study protocol. BMC Cancer. 2018 May 16;18(1):566. doi: 10.1186/s12885-018-4492-5. PMID 29769060